CLINICAL TRIAL: NCT05869123
Title: A Prospective Study to Evaluate Online Adaptive Radiotherapy in Postoperative Treatment of Endometrial and Cervical with Reduced Margin
Brief Title: Online Adaptive Radiotherapy for Postoperative Treatment of Endometrial and Cervical Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pumch-ART-1
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Uterine Cervical Neoplasm; Endometrial Neoplasms
Keywords: Uterine Cervical Neoplasm; Endometrial Neoplasms; Online Adaptive Radiotherapy; Adjuvant Radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Online Adaptive Radiotherapy (Experimental): Patients receive online adaptive radiotherapy with 5mm PTV margin. The CTV-N covered pelvic lymph nodes (common, internal and external iliac, obturator, and presacral) and CTV-V covered proximal vagina and any paravaginal or retracted parametrial tissue. A dose of 45 or 50.4Gy is delivered to CTV with online adaptive radiotherapy.
  Interventions: Radiation: Online adaptive radiotherapy

INTERVENTIONS:
Radiation: Online adaptive radiotherapy — PTV with 5 margins covers CTV

SUMMARY:
Online adaptive radiotherapy (oART) has demonstrated to be feasible to reduce planning target volume (PTV) margins for postoperative treatment of endometrial and cervical cancer. To explore the value of reduced margins in oART for postoperative treatment of endometrial and cervical cancer, we conducted a prospective clinical trial to determine the clinical efficacy and toxicity of reduced margins.

DETAILED DESCRIPTION:
This is an investigator-initiated efficacious, single-center, open-label clinical trial study. This study hypothesizes that the use of reduced PTV margins in oART for postoperative treatment of endometrial and cervical cancer could decrease toxicity and achieve more accurate dosimetric coverage. A dose of 45 or 50.4 Gy is delivered to clinical target volume (CTV) with reduced margin oART. Patients receive cisplatin based concurrent chemotherapy. The primary endpoint is acute toxicity. The first 10 patients were included in the study that have demonstrated the feasibility of reducing the margin (ClinicalTrials.gov ID: NCT05682950).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be informed of the investigational nature of this study and give written informed consent before treatment.
2. Postoperative endometrial and cervical cancer patients with pathologically confirmed no residual tumor at the resection margin and no evidence of distant metastasis (FIGO stage IVB).
3. Pathological findings indicate risk factors and adjuvant radiotherapy are prescribe.
4. Karnofsky score ≥ 70.
5. Subjects aged ≥ 18 years and ≤ 70 years.
6. No evidence of para-aortic metastatic lymph nodes.
7. No contraindications to CT scanning.
8. Subjects must be able to cooperate in completing the entire study.
9. Adequate marrow: neutrophile granulocyte count ≥1.5*10^9/L, hemoglobin ≥ 80 g/L, platelet count ≥100*10^9/L.
10. Normal liver and kidney function: Creatinine (Cr) < 1.5 mg/dl, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 2*upper limit of normal (ULN).

Exclusion Criteria:

1. Subjects who have received prior pelvic radiotherapy.
2. Subjects with other primary malignancies.
3. Subjects with contraindications to radiotherapy, as determined by the investigators.
4. Any severe disease which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control, and emotional disturbance.
5. Active infection with fever.
6. Active inflammatory bowel disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2025-03-03 (Estimated)

PRIMARY OUTCOMES:
Physician-reported acute toxicity | From the start of treatment to 3 months after treatment
  Physician-reported acute toxicity evaluated with Common Terminology Criteria for Adverse Events (CTCAE) 5.0

SECONDARY OUTCOMES:
Late toxicity evaluated with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme | 2-year
  Evaluated with Radiation Therapy Oncology Group (RTOG)/EORTC late radiation morbidity scoring scheme
The dose coverage of target volume as assessed by planing tumor volume V100% | Through study completion, an average of five month
  Planing tumor volume V100%, defined as the planing tumor volume receiving at least 100% of the prescribed dose (V100%), is used to evaluate the dose coverage of target volume.
Target automatically contouring accuracy | Through study completion, an average of five month
  For every target in each fraction, the evaluation of accuracy for target contouring are categorized as follow: no edits, minor edits, moderate edits, major edits and not applicable.
Organs at risk contouring accuracy | Through study completion, an average of five month
  For every organs at risk in each fraction, the evaluation of accuracy for organs at risk contouring are categorized as follows: no edits, minor edits, moderate edits, major edits and not applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Fuquan Zhang, M.D., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Jong R, Visser J, van Wieringen N, Wiersma J, Geijsen D, Bel A. Feasibility of Conebeam CT-based online adaptive radiotherapy for neoadjuvant treatment of rectal cancer. Radiat Oncol. 2021 Jul 23;16(1):136. doi: 10.1186/s13014-021-01866-7. PMID 34301300
- [Background] Schiff JP, Stowe HB, Price A, Laugeman E, Hatscher C, Hugo GD, Badiyan SN, Kim H, Robinson CG, Henke LE. In Silico Trial of Computed Tomography-Guided Stereotactic Adaptive Radiation Therapy (CT-STAR) for the Treatment of Abdominal Oligometastases. Int J Radiat Oncol Biol Phys. 2022 Dec 1;114(5):1022-1031. doi: 10.1016/j.ijrobp.2022.06.078. Epub 2022 Jun 26. PMID 35768023